CLINICAL TRIAL: NCT04919148
Title: Climate Change Beliefs, Perceived Risk of Heat Stress and Responses to Heat Health Warnings Among the General Public of Hong Kong: a Mixed-methods Study
Brief Title: Perceptions of Weather Risks and Climate Beliefs Among the Hong Kong General Public
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Qiuyan Liao, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: UW 19-093
Record Dates: First submitted 2021-05-28; First posted 2021-06-09 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Weather Risk Perception

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants receive control message (No Intervention): Participants only receive standard heat risk warning
- Participants receive intervention message (Experimental): Participants receive standard heat risk warning plus figures incorporating the health impacts of heat and pro-environment behaviors.
  Interventions: Behavioral: Heat risk and pro-environment behavior message

INTERVENTIONS:
Behavioral: Heat risk and pro-environment behavior message — Eligible participants will be randomized to either a control condition to receive a standardized heat health warning or an intervention condition to receive a heat health warning plus figures depicting heat risk and pro-environment behavior via their preferred and accessible channel (WhatsApp, WeChat or the text message) each time when a Very Hot Weather Warning is issued by the Hong Kong Observatory.
  Arms: Participants receive intervention message

SUMMARY:
Background: Local abnormal heat events may be used as proxies for communicating the health impacts of climate change when people physically feel the effects to reduce the psychological distance of climate change and improve public engagement with climate and weather risk. However, there are concerns that this strategy may be more effective for climate believers, and that it may somewhat compromise the scientific precision because it may lead to erroneous beliefs that climate change is merely characterized by temperature rises or extreme heat but ignore other extreme weather events such as flood and extreme cold, and that cold spells are interpreted as evidence of no climate change. None of these potential effects and concerns has been tested.

Aims: This proposed study is aimed to explore patterns of climate beliefs and their influences on perceptions of heat-related risks and responses to heat health warnings in the general public of Hong Kong; (2) Test the preliminary effects of a revised heat health warning (RHHW) that incorporates information about the health impacts of climate change into existing heat health warning on perceived heat-related risk and climate beliefs.

Design and subjects: This will be a mix-methods study comprising in-depth qualitative interviews, a population-based cohort survey and a pilot randomized control trial (RCT). Subjects will be the general Hong Kong Chinese adults aged ≥18 years.

Main outcome measures: Latent class analysis will be conducted to examine patterns of climate beliefs while structural equation modelling to test the relationships among climate beliefs, perceived heat-related risks and behavioural responses to heat warnings. Qualitative data will be analysed using thematic content analysis while the effect of RHHW will be tested using t-test and linear regression models.

ELIGIBILITY:
Inclusion Criteria:

* Participants should own a mobile phone and be able to read Chinese.

Exclusion Criteria:

* Participants with no mobile phone or cannot understand Chinese will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 429 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Emotional engagement with heat and climate change risk (emotional valence) | One week after completion of all messages delivery
  Measure participants' emotional engagement with risk of heat stress and climate change, in specific, participants will be asked to indicate how they feel about the health impacts of climate change (using a slider from -3 to 3). Higher scores indicate more positive emotion.
Emotional engagement with heat and climate change risk (discrete emotion) | One week after completion of all messages delivery
  Participants will be asked how much they feel fear/helpless/worried/disgust when thinking about health impacts of climate change (on a 7-point Likert scale). Higher scores indicate stronger emotion arousal.
Short-term effect of risk perception toward heat and climate change risk | One week after completion of all messages delivery
  Their perceived health risk toward climate change and heat stress will be measured using items derived from our baseline and follow-up surveys (likelihood, severity and perceived worry will be used to gauge participants' risk perception). All measures on a 5-point likert scale with higher scores indicating greater risk perception.
Long-term effect of risk perception toward heat and climate change | One month after completion of all messages delivery
  Their perceived health risk toward climate change and heat stress will be measured using items derived from our baseline and follow-up surveys (likelihood, severity and perceived worry will be used to gauge participants' risk perception). All measures on a 5-point likert scale with higher scores indicating greater risk perception.

SECONDARY OUTCOMES:
Short-term effect of self-efficacy in taking pro-environment actions | One week after completion of all messages delivery
  Perceived self-efficacy in taking actions to mitigate climate change will be measured by four items derived from previous baseline and follow-up surveys.(Items include: 1) I can personally help to reduce climate change by changing my behavior 2) There are a variety of external factors that make it difficult for me to take actions that help to reduce climate change 3) My action to reduce the effects of climate change in my community will encourage others to reduce the effect of climate change through their own actions 4) If I want, it is easy for me to take actions to help tackle climate change). Responses will be rated on a 5-point Likert (Strongly disagree/Disagree/Agree/Strongly agree/No opinion).
Long-term effect of self-efficacy in taking pro-environment actions | One month after completion of all messages delivery
  Perceived self-efficacy in taking actions to mitigate climate change will be measured by four items derived from previous baseline and follow-up surveys.(Items include: 1) I can personally help to reduce climate change by changing my behavior 2) There are a variety of external factors that make it difficult for me to take actions that help to reduce climate change 3) My action to reduce the effects of climate change in my community will encourage others to reduce the effect of climate change through their own actions 4) If I want, it is easy for me to take actions to help tackle climate change). Responses will be rated on a 5-point Likert (Strongly disagree/Disagree/Agree/Strongly agree/No opinion).
Short-term effect of intention in taking pro-environment actions | One week after completion of all messages delivery
  Participants will also be asked to indicate their intention to 1) reduce energy waste 2) buy energy efficient products, and 3) change some of the daily habits to help tackle climate change. Responses will be rated on a 7-point Likert scale. Higher scores indicate greater behavioral intention.
Long-term effect of intention in taking pro-environment actions | One month after completion of all messages delivery
  Participants will also be asked to indicate their intention to 1) reduce energy waste 2) buy energy efficient products, and 3) change some of the daily habits to help tackle climate change. Responses will be rated on a 7-point Likert scale. Higher scores indicate greater behavioral intention.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hong Kong School of Public Health, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
Derived data supporting the findings of this study are available from the corresponding author on reasonable request.